CLINICAL TRIAL: NCT05223023
Title: Opinions of Physiotherapists Working in the Area of Pediatric Rehabilitation About Treatment Types, Effectiveness and Training
Brief Title: Opinions of Physiotherapists Working in the Area of Pediatric Rehabilitation
Acronym: physio
Status: Completed | Type: Observational
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, Hatice Adiguzel, Assistant Proffessor, Kahramanmaras Sutcu Imam University
Other Study IDs: KSUFTR3
Record Dates: First submitted 2022-01-24; First posted 2022-02-03 (Actual); Last update posted 2022-02-18 (Actual); Status verified 2022-02

CONDITIONS: Pediatric ALL; Physician's Role; Educational Problems; Occupational Problems
Keywords: awareness; physical therapists; pediatric rehabilitation; treatment types; opinion; physiotherapy; training
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1/Assessment of the opinions of the physiotherapists: All of the therapists who works in the pediatric rehabilitation area were assessed with the scale of 50 questions named "Opinions of Physiotherapists Working in the Area of Pediatric Rehabilitation on Treatment Types, Efficiency and Training"
  Interventions: Other: questionnaire

INTERVENTIONS:
Other: questionnaire — All of the therapists who works in the pediatric rehabilitation area were assessed with the scale of 50 questions named "Opinions of Physiotherapists Working in the Area of Pediatric Rehabilitation on Treatment Types, Efficiency and Training"
  Other Names: assesments of the physiotherapists opinions who works in the area of pediatric rehabilitation

SUMMARY:
According to the definition of the World Confederation of Physical Therapy (WCPT), physiotherapists serve to restore, maintain and improve the movement and functional skills of individuals. Physiotherapists; They take a role when the movement and functions of people are endangered due to aging, injury, disease, disorder or environmental factors. As in the world, the physiotherapist profession is gradually developing and spreading in Turkey. In this sense, the number of Physiotherapy and Rehabilitation faculties, departments and colleges is increasing every year. With the increasing prevalence of the profession, it has brought up the revision of training programs and questioning their success. In the literature, there are accreditation reports and guides in Australia, America and Canada regarding the education of the Physiotherapy and Rehabilitation science field. When we look at the literature in our country, there is no study that covers a common curriculum or training program developed for Physiotherapy and Rehabilitation in Turkey.Therefore, it is thought that the diversity in education programs may affect the way physiotherapists, most of whom work in special education, work after graduation.

DETAILED DESCRIPTION:
In a study evaluating how the employment period and employment status of physiotherapists who graduated in the 2012-2016 period are affected; it was determined that pediatric rehabilitation is the area where physiotherapists work the most with a rate of 44.6%. In another study, it was stated that according to the managers of special education and rehabilitation centers, different branches working in these institutions should reflect their knowledge of special education. However, it has been stated that the personnel employed in the special education and rehabilitation centers opened to serve children with disabilities generally do not have sufficient knowledge and formation about the education and rehabilitation of individuals who need special education.

In the process of increasing awareness, which forms the basis of development, which is a cognitive and sensory activity, the individual perceives the life in which he lives in relation to his feelings, wishes, dreams and behaviors. Increasing the level of awareness enables the individual to enrich his/her way of reacting to the situations he/she experiences and to discover different methods in his/her relationships and life, thanks to some new cognitive schemas formed in the mind. Professional awareness provides preliminary information on concepts such as the competencies of that profession, the groups they are in contact with, the laws and regulations related to the profession, duties and responsibilities, the individual's psychological and physical suitability for the profession, and professional sensitivity. Formation of professional awareness in physiotherapists; In case of all kinds of injuries, illnesses and disabilities that cause movement disorders, reintegration of individuals with physical disabilities in workplace health and industry, development of the concept of rehabilitation, which has an important role in preventive health services for healthy individuals and in increasing the quality of life, increasing the quality of health services, illness It is very important in terms of achieving professional goals that will affect the whole society, such as minimizing disability and disability. When the studies on this subject in Turkey in the organization named "European Network of Physiotherapy in Higher Education" are examined, it is seen that awareness trainings are not included in the physiotherapy profession.The aim of this study, which is planned with these predictions; To determine the professional awareness levels of physiotherapists working in the areo of pediatric rehabilitation. It is thought that this study can be a guide in terms of determining the aims and qualifications of physiotherapists, revealing professional requirements, developing new curriculum and awareness training programs, determining the subjects on which training programs should be conducted, and thus raising more beneficial professionals to the society.

ELIGIBILITY:
Inclusion Criteria:

* Physiotherapists between the ages of 22-50 who are actively working in the area of pediatric rehabilitation and participating in the study voluntarily

Exclusion Criteria:

* Therapists who were not willing to answer the questionnaire

Ages: 22 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Physiotherapists between the ages of 22-50 who are actively working in the area of pediatric rehabilitation and participating in the study voluntarily
Sampling Method: Non-Probability Sample
Enrollment: 83 (Actual)
Dates: Start 2019-04-30 (Actual); Primary Completion 2019-06-15 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
The questionnaire of the Opinions of Physiotherapists Working in the Area of Pediatric Rehabilitation on Treatment Types, Efficiency and Training | first day of assessment
  All of the therapists who works in the pediatric rehabilitation area were assessed with the scale of 50 questions named "Opinions of Physiotherapists Working in the Area of Pediatric Rehabilitation on Treatment Types, Efficiency and Training". Both multiple choice and open-ended answers are marked in the questionnaire. The questionnaire provides insight into all therapeutic practices and uses of therapy diversity. The survey was prepared by the researchers. There is no specific score range. But there will be 2 or 3 true answers in each question. Also there will be some wrong answers in some questions. True and false answer will be shown in frequency and % in data analysis.

SECONDARY OUTCOMES:
Physiotherapists' gender | first day of assessment
  Physiotherapists gender was recoorded as male, female.
Physiotherapists' weight | first day of assessment
  Physiotherapists' weight was recoorded as kilograms.
Physiotherapists' length | first day of assessment
  Physiotherapists' length was recoorded as centimeter (cm)
Physiotherapists' occupation year | first day of assessment
  Physiotherapists' occupation year was recorded as year.
Physiotherapists' graduation year | first day of assessment
  Physiotherapists' graduation year was recorded as year.
Education level of physiotherapists | first day of assessment
  Education level of physiotherapists was recordes as licence, master or PHD.

CONTACTS AND LOCATIONS:
Overall Officials: hatice adıgüzel, PhD, Principal Investigator — Kahramanmaras Sutcu Imam University; Nevin Ergun, Proffessor, Study Director — Sanko University
Locations (1):
- Kahramanmaras Sutcu Imam University, Kahramanmaraş, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No